CLINICAL TRIAL: NCT06799559
Title: A Multicenter, Randomized, Double-blind, Parallel Controlled Study on the Efficacy and Safety of QLM1016 in the Treatment of Schizophrenia
Brief Title: Study on the Efficacy and Safety of QLM1016 in Schizophrenia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLM1016-301
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLM1016 (Experimental)
  Interventions: Drug: 3-6mg QLM1016
- Aripiprazole oral solution film (Active Comparator)
  Interventions: Drug: 10-20 mg Aripiprazole oral solution film

INTERVENTIONS:
Drug: 3-6mg QLM1016 — 3-6mg QLM1016 pluse Aripiprazole dummy oral solution film administered orally once daily for 6 weeks
  Arms: QLM1016
Drug: 10-20 mg Aripiprazole oral solution film — 10-20mg Aripiprazole oral solution film plus QLM1016 dummy oral solution film administered orally once daily for 6 weeks.
  Arms: Aripiprazole oral solution film

SUMMARY:
The study will evaluate the antipsychotic efficacy of QLM1016 in a multicenter, randomized, double-blind, parallel controlled study in patients diagnosed with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects, ages 18-65 inclusive, with a clinical diagnosis of schizophrenia
* PANSS total score ≥ 70 and ≤ 120，Rating of at least 4 (moderate) on at least 2 of the following 4 PANSS positive symptoms: delusions, hallucinatory behavior, conceptual disorganization, and unusual thought content
* CGI-S score ≥ 4

Exclusion Criteria:

* Currently, meet DSM-5 diagnostic criteria for other psychiatric disorders ( for example schizoaffective disorder, schizophreniform disorder, bipolar I and II disorder; pervasive developmental disorder, mental retardation, delirium, dementia, amnestic and other cognitive disorders；
* known or suspected borderline or antisocial personality disorder or other psychiatric disorders of sufficient severity to interfere with participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline to week 6 in the Positive and Negative Syndrome Scale (PANSS) total score | Time Frame: 6 weeks